CLINICAL TRIAL: NCT03482453
Title: Phase 1, Randomized, Double-blind, Placebo-Controlled, Single Rising Dose Study to Evaluate Pharmacokinetics, Safety, and Tolerability of TAK-788 Followed by Open-Label, Crossover Evaluation of the Effects of a Low-Fat Meal on TAK-788 Pharmacokinetics and Evaluation of Relative Bioavailability of TAK-788 Capsules in Healthy Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics (PK), Safety and Tolerability of TAK-788 Followed by Evaluation of the Effects of a Low-Fat Meal on TAK-788 PK and Evaluation of Relative Bioavailability of TAK-788 Capsules in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: TAK-788-1001; U1111-1208-9582 (Other: WHO)
Record Dates: First submitted 2018-03-23; First posted 2018-03-29 (Actual); Results first posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — mobocertinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1 Cohort 1: TAK-788 (Experimental): TAK-788, capsule, orally or TAK-788 matching placebo capsule, orally, once under fasted conditions on Day 1.
  Interventions: Drug: TAK-788; Drug: Placebo
- Part 1 Cohort 2: TAK-788 (Experimental): TAK-788, capsule, orally or TAK-788 matching placebo capsule, orally, once under fasted conditions on Day 1 following review of safety data from Cohort 1.
  Interventions: Drug: TAK-788; Drug: Placebo
- Part 1 Cohort 3: TAK-788 (Experimental): TAK-788, capsule, orally or TAK-788 matching placebo capsule, orally, once under fasted conditions on Day 1 following review of safety data from Cohort 2.
  Interventions: Drug: TAK-788; Drug: Placebo
- Part 1 Cohort 4: TAK-788 (Experimental): TAK-788, capsule, orally or TAK-788 matching placebo capsule, orally, once under fasted conditions on Day 1 following review of safety data from Cohort 3.
  Interventions: Drug: TAK-788; Drug: Placebo
- Part 1 Cohort 5: TAK-788 (Experimental): TAK-788, capsule, orally or TAK-788 matching placebo capsule, orally, once under fasted conditions on Day 1 following review of safety data from Cohort 4.
  Interventions: Drug: TAK-788; Drug: Placebo
- Part 2: TAK-788 Fed + TAK-788 Fasted (Experimental): TAK-788, capsule, orally, once on Day 1 of Intervention Period 1 under fed conditions with low-fat meal (Treatment A), followed by at least 7 days washout period, further followed by TAK-788, capsule, orally, once on Day 1 of Intervention Period 2 under fasted conditions (Treatment B). TAK-788 dose will be determined based on review of safety and tolerability data from cohorts of Part 1.
  Interventions: Drug: TAK-788
- Part 2: TAK-788 Fasted + TAK-788 Fed (Experimental): TAK-788, capsule, orally, once on Day 1 of Intervention Period 1 under fasted conditions (Treatment B), followed by at least 7 days washout period, further followed by TAK-788, capsule, orally, once on Day 1 of Intervention Period 2 under fed conditions with low-fat meal (Treatment A). TAK-788 dose will be determined based on review of safety and tolerability data from cohorts of Part 1.
  Interventions: Drug: TAK-788
- Part 3: TAK-788 DiC (reference) + TAK-788 DiC (test) (Experimental): TAK-788 160 mg, DiC A (reference), orally, under fasted condition, once on Day 1 of Intervention Period 1, followed by at least 7 days washout period, further followed by TAK-788 160 mg, DiC B (test), orally, under fasted condition, once on Day 1 of Intervention Period 2.
  Interventions: Drug: TAK-788
- Part 3: TAK-788 DiC (test) + TAK-788 DiC (reference) (Experimental): TAK-788 160 mg, DiC B (test), orally, under fasted condition, once, on Day 1 of Intervention Period 1, followed by at least 7 days washout period, further followed by TAK-788 160 mg, DiC A (reference), orally, under fasted condition, once on Day 1 of Intervention Period 2.
  Interventions: Drug: TAK-788

INTERVENTIONS:
Drug: TAK-788 — TAK-788 capsules.
  Other Names: AP32788
  Arms: Part 1 Cohort 1: TAK-788; Part 1 Cohort 2: TAK-788; Part 1 Cohort 3: TAK-788; Part 1 Cohort 4: TAK-788; Part 1 Cohort 5: TAK-788; Part 2: TAK-788 Fasted + TAK-788 Fed; Part 2: TAK-788 Fed + TAK-788 Fasted
Drug: Placebo — TAK-788 placebo-matching capsules.
  Arms: Part 1 Cohort 1: TAK-788; Part 1 Cohort 2: TAK-788; Part 1 Cohort 3: TAK-788; Part 1 Cohort 4: TAK-788; Part 1 Cohort 5: TAK-788
Drug: TAK-788 — TAK-788 DiC.
  Other Names: AP32788
  Arms: Part 3: TAK-788 DiC (reference) + TAK-788 DiC (test); Part 3: TAK-788 DiC (test) + TAK-788 DiC (reference)

SUMMARY:
The purpose of this study is to assess the safety, tolerability of TAK-788 and to identify a tolerable single oral dose of TAK-788 administered as a drug-in-capsule (DiC) formulation, to characterize the effects of a low-fat meal on the PK of the TAK-788 administered as DiC formulation and to evaluate the bioavailability of a test (Process B) DiC of TAK-788 relative to a reference (Process A) DiC of TAK-788 in healthy participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-788. The study will assess the safety and tolerability of single oral dose of TAK-788, evaluate the effect of a low-fat meal on PK of TAK-788 and will assess the relative bioavailability of two DiCs of TAK-788.

The study will enroll approximately 69 participants. The study is designed to consist of 3 parts: Part 1- dose escalation phase, Part 2- low fat meal effect and Part 3 - relative bioavailability. The study population of Part 1 will consist of 40 participants enrolled into 5 cohorts. Each cohort will have 8 randomized participants with 6 receiving a single dose of TAK-788, and 2 receiving matching placebo under fasted conditions. In Cohorts 1 to 5, safety of single-dose TAK-788 will be evaluated. For Part 2, the effect of a low-fat meal on a single tolerable dose of TAK-788 will be determined following review of safety and tolerability data from the previous cohorts in Part 1. The study population of Part 2 will consist of 16 participants enrolled into 2 cohorts of different doses, where participants will be randomized to a cross-over sequence of:

* TAK-788 Fed + TAK-788 Fasted
* TAK-788 Fasted + TAK-788 Fed

The study population of Part 3 will consist of 13 participants enrolled into 1 cohort, where participants will be randomized to a cross-over sequence of:

* TAK-788 DiC (reference) + TAK-788 DiC (test)
* TAK-788 DiC (test) + TAK-788 DiC (reference) This single-center trial will be conducted in the United States. The overall time to participate in this study is approximately 7 months. Participants will be contacted by telephone 30 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Body weight of greater than or equal to (>=) 45 kilogram (kg) (women) or >=55 kg (men) and a body mass index of 18.0 to 30.0 kilogram per square meter (kg/m^2) at screening.
2. Nonsmoker (never smoked or greater than [>] 20 years from last occurrence of smoking).
3. Normal organ function including hepatic, renal, and bone marrow function.

Exclusion Criteria:

1. Manifestations of malabsorption due to prior gastro-intestinal (GI) surgery, GI disease, or for an unknown other reason that may alter the PK of TAK-788.
2. Pulmonary infection ongoing or within 30 days of informed consent.
3. Inability to undergo venipuncture and/or tolerate venous access.
4. Inability to tolerate multiple blood sampling.
5. Ongoing or active infection, including but not limited to, the requirement for intravenous (IV) antibiotics.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2018-12-22 (Actual); Study Completion 2019-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- PRA Health Sciences, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 28 March 2018 to 18 January 2019.
Pre-assignment Details: Healthy participants were enrolled in this 3 parts study to receive: TAK-788 as a single rising dose of 20 milligram (mg), 40 mg, 80 mg, 120 mg, 160 mg in Part 1; TAK-788 in a 2-way cross-over design with or without a low-fat meal in Part B; or in a 2-way cross-over sequence to receive TAK-788 drug in capsule (DiC) A or B in Part 3.
Groups:
- Part 1: Pooled Placebo: TAK-788 matching placebo capsule, orally, once under fasted conditions on Day 1.
- Part 1 Cohort 1: TAK-788 20 mg: TAK-788 20 mg, capsule, orally, once under fasted conditions on Day 1.
- Part 1 Cohort 2: TAK-788 40 mg: TAK-788 40 mg, capsule, orally, once under fasted conditions on Day 1.
- Part 1 Cohort 3: TAK-788 80 mg: TAK-788 80 mg, capsule, orally, once under fasted conditions on Day 1.
- Part 1 Cohort 4: TAK-788 120 mg: TAK-788 120 mg, capsule, orally, once under fasted conditions on Day 1.
- Part 1 Cohort 5: TAK-788 160 mg: TAK-788 160 mg, capsule, orally, once under fasted conditions on Day 1.
- Part 2: TAK-788 120 mg Fed + TAK-788 120 mg Fasted: TAK-788 120 mg, capsule, orally, once on Day 1 of Intervention Period 1 under fed conditions with low-fat meal (Treatment A), followed by at least 7 days washout period, further followed by TAK-788, 120 mg, capsule, orally, once on Day 1 of Intervention Period 2 under fasted conditions (Treatment B).
- Part 2: TAK-788 120 mg Fasted + TAK-788 120 mg Fed: TAK-788, 120 mg, capsule, orally, once on Day 1 of Intervention Period 1 under fasted conditions (Treatment B), followed by at least 7 days washout period, further followed by TAK-788, 120 mg, capsule, orally, once on Day 1 of Intervention Period 2 under fed conditions with low-fat meal (Treatment A).
- Part 2: TAK-788 160 mg Fed + TAK-788 160 mg Fasted: TAK-788 160 mg, capsule, orally, once on Day 1 of Intervention Period 1 under fed conditions with low-fat meal (Treatment A), followed by at least 7 days washout period, further followed by TAK-788 160 mg, capsule, orally, once on Day 1 of Intervention Period 2 under fasted conditions (Treatment B).
- Part 2: TAK-788 160 mg Fasted + TAK-788 160 mg Fed: TAK-788, 160 mg, capsule, orally, once on Day 1 of Intervention Period 1 under fasted conditions (Treatment B), followed by at least 7 days washout period, further followed by TAK-788, 160 mg, capsule, orally, once on Day 1 of Intervention Period 2 under fed conditions with low-fat meal (Treatment A).
- Part 3: TAK-788 DiC A + TAK-788 DiC B: TAK-7 160 mg, DiC A (reference), orally, under fasted condition, once on Day 1 of Intervention Period 1, followed by at least 7 days washout period, further followed by TAK-788 160 mg, DiC B (test), orally, under fasted condition, once on Day 1 of Intervention Period 2.
- Part 3: TAK-788 DiC B + TAK-788 DiC A: TAK-788 160 mg, DiC B (test), orally, under fasted condition, once on Day 1 of Intervention Period 1, followed by at least 7 days washout period, further followed by TAK-788 160 mg, DiC A (reference), orally, under fasted condition, once on Day 1 of Intervention Period 2.
Period: Part 1 (1 Day)
Arm/Group | Part 1: Pooled Placebo | Part 1 Cohort 1: TAK-788 20 mg | Part 1 Cohort 2: TAK-788 40 mg | Part 1 Cohort 3: TAK-788 80 mg | Part 1 Cohort 4: TAK-788 120 mg | Part 1 Cohort 5: TAK-788 160 mg | Part 2: TAK-788 120 mg Fed + TAK-788 120 mg Fasted | Part 2: TAK-788 120 mg Fasted + TAK-788 120 mg Fed | Part 2: TAK-788 160 mg Fed + TAK-788 160 mg Fasted | Part 2: TAK-788 160 mg Fasted + TAK-788 160 mg Fed | Part 3: TAK-788 DiC A + TAK-788 DiC B | Part 3: TAK-788 DiC B + TAK-788 DiC A
Started | 10 | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 10 | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Parts 2, 3 Intervention Period 1 (1 Day)
Arm/Group | Part 1: Pooled Placebo | Part 1 Cohort 1: TAK-788 20 mg | Part 1 Cohort 2: TAK-788 40 mg | Part 1 Cohort 3: TAK-788 80 mg | Part 1 Cohort 4: TAK-788 120 mg | Part 1 Cohort 5: TAK-788 160 mg | Part 2: TAK-788 120 mg Fed + TAK-788 120 mg Fasted | Part 2: TAK-788 120 mg Fasted + TAK-788 120 mg Fed | Part 2: TAK-788 160 mg Fed + TAK-788 160 mg Fasted | Part 2: TAK-788 160 mg Fasted + TAK-788 160 mg Fed | Part 3: TAK-788 DiC A + TAK-788 DiC B | Part 3: TAK-788 DiC B + TAK-788 DiC A
Started | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 5 | 5 | 7 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 5 | 5 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Parts 2, 3 Washout Period (7 Days)
Arm/Group | Part 1: Pooled Placebo | Part 1 Cohort 1: TAK-788 20 mg | Part 1 Cohort 2: TAK-788 40 mg | Part 1 Cohort 3: TAK-788 80 mg | Part 1 Cohort 4: TAK-788 120 mg | Part 1 Cohort 5: TAK-788 160 mg | Part 2: TAK-788 120 mg Fed + TAK-788 120 mg Fasted | Part 2: TAK-788 120 mg Fasted + TAK-788 120 mg Fed | Part 2: TAK-788 160 mg Fed + TAK-788 160 mg Fasted | Part 2: TAK-788 160 mg Fasted + TAK-788 160 mg Fed | Part 3: TAK-788 DiC A + TAK-788 DiC B | Part 3: TAK-788 DiC B + TAK-788 DiC A
Started | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 5 | 5 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 5 | 5 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Parts 2, 3 Intervention Period 2 (1 Day)
Arm/Group | Part 1: Pooled Placebo | Part 1 Cohort 1: TAK-788 20 mg | Part 1 Cohort 2: TAK-788 40 mg | Part 1 Cohort 3: TAK-788 80 mg | Part 1 Cohort 4: TAK-788 120 mg | Part 1 Cohort 5: TAK-788 160 mg | Part 2: TAK-788 120 mg Fed + TAK-788 120 mg Fasted | Part 2: TAK-788 120 mg Fasted + TAK-788 120 mg Fed | Part 2: TAK-788 160 mg Fed + TAK-788 160 mg Fasted | Part 2: TAK-788 160 mg Fasted + TAK-788 160 mg Fed | Part 3: TAK-788 DiC A + TAK-788 DiC B | Part 3: TAK-788 DiC B + TAK-788 DiC A
Started | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 5 | 5 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 5 | 5 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all participants who received any study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Pooled Placebo | Part 1 Cohort 1: TAK-788 20 mg | Part 1 Cohort 2: TAK-788 40 mg | Part 1 Cohort 3: TAK-788 80 mg | Part 1 Cohort 4: TAK-788 120 mg | Part 1 Cohort 5: TAK-788 160 mg | Part 2: TAK-788 120 mg Fed + TAK-788 120 mg Fasted | Part 2: TAK-788 120 mg Fasted + TAK-788 120 mg Fed | Part 2: TAK-788 160 mg Fed + TAK-788 160 mg Fasted | Part 2: TAK-788 160 mg Fasted + TAK-788 160 mg Fed | Part 3: TAK-788 DiC A + TAK-788 DiC B | Part 3: TAK-788 DiC B + TAK-788 DiC A | Total
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 3 | 3 | 5 | 5 | 7 | 6 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 6 | 6 | 6 | 6 | 6 | 3 | 3 | 5 | 5 | 7 | 6 | 69
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 1 | 2 | 3 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 17
  Male | 7 | 6 | 5 | 4 | 3 | 5 | 2 | 2 | 4 | 4 | 5 | 5 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 10
  Not Hispanic or Latino | 9 | 5 | 5 | 5 | 5 | 6 | 3 | 3 | 4 | 5 | 5 | 4 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
  White | 9 | 6 | 6 | 6 | 6 | 6 | 3 | 3 | 5 | 4 | 7 | 5 | 66
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 6 | 6 | 6 | 6 | 6 | 3 | 3 | 5 | 5 | 7 | 6 | 69

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Time Frame: Baseline up to 30 days after the last dose of study drug (Day 31)
Population: The safety set included all participants who received any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Pooled Placebo | Part 1 Cohort 1: TAK-788 20 mg | Part 1 Cohort 2: TAK-788 40 mg | Part 1 Cohort 3: TAK-788 80 mg | Part 1 Cohort 4: TAK-788 120 mg | Part 1 Cohort 5: TAK-788 160 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Participants | 2 | 2 | 3 | 4 | 3 | 5

2. Primary Outcome: Part 1: Number of Participants With One or More Serious Adverse Events (SAEs)
Time Frame: Baseline up to 30 days after the last dose of study drug (Day 31)
Population: The safety set included all participants who received any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Pooled Placebo | Part 1 Cohort 1: TAK-788 20 mg | Part 1 Cohort 2: TAK-788 40 mg | Part 1 Cohort 3: TAK-788 80 mg | Part 1 Cohort 4: TAK-788 120 mg | Part 1 Cohort 5: TAK-788 160 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Part 1: Number of Participants With Clinically Significant Abnormal Laboratory Values
Time Frame: Baseline up to 30 days after the last dose of study drug (Day 31)
Population: The safety set included all participants who received any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Pooled Placebo | Part 1 Cohort 1: TAK-788 20 mg | Part 1 Cohort 2: TAK-788 40 mg | Part 1 Cohort 3: TAK-788 80 mg | Part 1 Cohort 4: TAK-788 120 mg | Part 1 Cohort 5: TAK-788 160 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part 1: Number of Participants With Clinically Significant Abnormal Vital Signs
Time Frame: Baseline up to 30 days after the last dose of study drug (Day 31)
Population: The safety set included all participants who received any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Pooled Placebo | Part 1 Cohort 1: TAK-788 20 mg | Part 1 Cohort 2: TAK-788 40 mg | Part 1 Cohort 3: TAK-788 80 mg | Part 1 Cohort 4: TAK-788 120 mg | Part 1 Cohort 5: TAK-788 160 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Part 2, Cmax: Maximum Observed Plasma Concentration for TAK-788
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: The pharmacokinetic (PK) set included all participants in the safety set who had no major protocol deviations that would have affected the PK analysis and who had sufficient data to calculate PK parameters.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- Part 2: TAK-788 120 mg Fed: TAK-788 120 mg, capsule, orally, under fed conditions with low-fat meal (Treatment A), once on Day 1 of either Intervention Period 1 or 2.
- Part 2: TAK-788 120 mg Fasted: TAK-788, 120 mg, capsule, orally, under fasted conditions (Treatment B), once on Day 1 of either Intervention Period 1 or 2.
- Part 2: TAK-788 160 mg Fed: TAK-788, 160 mg, capsule, orally, under fed conditions with low-fat meal (Treatment A), once on Day 1 of either Intervention Period 1 or 2.
- Part 2: TAK-788 160 mg Fasted: TAK-788, 160 mg, capsule, orally, under fasted conditions (Treatment B), once on Day 1 of either Intervention Period 1 or 2.
Arm/Group | Part 2: TAK-788 120 mg Fed | Part 2: TAK-788 120 mg Fasted | Part 2: TAK-788 160 mg Fed | Part 2: TAK-788 160 mg Fasted
Number analyzed (Participants) | 6 | 6 | 10 | 10
nanogram per milliliter (ng/mL) | 27.52 (11.423) | 31.24 (16.682) | 39.51 (17.179) | 41.00 (21.917)
Statistical Analysis 1: Comparison: Part 2: TAK-788 120 mg Fed vs Part 2: TAK-788 120 mg Fasted; Test type: Equivalence — A linear mixed effect model on the natural log-transformed parameters was performed with regimen, sequence and period as a fixed effect and subject nested within sequence as a random effect. The least square means (LS means) for the log-transformed parameters were exponentiated to obtain the point estimates and 90 percent (%) Confidence Intervals (CIs) of the geometric LS mean ratio on the original scale; Geometric LS Mean Ratio = 0.8810, 90% CI 2-sided [0.7108 to 1.0921]
Statistical Analysis 2: Comparison: Part 2: TAK-788 160 mg Fed vs Part 2: TAK-788 160 mg Fasted; Test type: Equivalence — A linear mixed effect model on the natural log-transformed parameters was performed with regimen, sequence and period as a fixed effect and subject nested within sequence as a random effect. The LS means for the log-transformed parameters were exponentiated to obtain the point estimates and 90% CIs of the geometric LS mean ratio on the original scale; Geometric LS Mean Ratio = 0.9637, 90% CI 2-sided [0.8361 to 1.1107]

6. Primary Outcome: Part 3, Cmax: Maximum Observed Plasma Concentration for TAK-788
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: The PK set included all participants in the safety set who had no major protocol deviations that would have affected the PK analysis and who had sufficient data to calculate PK parameters.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Groups:
- Part 3: TAK-788 DiC A: TAK-788 160 mg, DiC A (reference), orally, under fasted condition, once on Day 1 of either Intervention Period 1 or 2.
- Part 3: TAK-788 DiC B: TAK-788 160 mg, DiC B (test), orally, under fasted condition, once on Day 1 of either Intervention Period 1 or 2.
Arm/Group | Part 3: TAK-788 DiC A | Part 3: TAK-788 DiC B
Number analyzed (Participants) | 12 | 12
ng/mL | 44.77 (14.738) | 41.71 (11.931)
Statistical Analysis 1: Comparison: Part 3: TAK-788 DiC A vs Part 3: TAK-788 DiC B; Test type: Equivalence — [test comment as in outcome 5, analysis 2]; Geometric LS Mean Ratio = 0.9317, 90% CI 2-sided [0.8458 to 1.0263]

7. Primary Outcome: Part 2, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-788
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hour
Arm/Group | Part 2: TAK-788 120 mg Fed | Part 2: TAK-788 120 mg Fasted | Part 2: TAK-788 160 mg Fed | Part 2: TAK-788 160 mg Fasted
Number analyzed (Participants) | 6 | 6 | 10 | 10
hour | 6.0 [4 to 8] | 4.0 [2 to 6] | 6.0 [2 to 8] | 6.0 [2 to 12]

8. Primary Outcome: Part 3, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-788
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hour
Arm/Group | Part 3: TAK-788 DiC A | Part 3: TAK-788 DiC B
Number analyzed (Participants) | 12 | 12
hour | 6.0 [2 to 8] | 5.0 [2 to 8]

9. Primary Outcome: Part 2, AUCt: Area Under the Plasma Concentration-time Curve From Time 0 to Time t for TAK-788
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Part 2: TAK-788 120 mg Fed | Part 2: TAK-788 120 mg Fasted | Part 2: TAK-788 160 mg Fed | Part 2: TAK-788 160 mg Fasted
Number analyzed (Participants) | 6 | 6 | 10 | 10
hour*nanogram per milliliter (h*ng/mL) | 526.3 (272.72) | 518.3 (300.84) | 700.6 (295.10) | 733.6 (461.41)

10. Primary Outcome: Part 3, AUCt: Area Under the Plasma Concentration-time Curve From Time 0 to Time t for TAK-788
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 3: TAK-788 DiC A | Part 3: TAK-788 DiC B
Number analyzed (Participants) | 12 | 12
h*ng/mL | 706.1 (173.63) | 677.9 (239.28)

11. Primary Outcome: Part 2, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-788
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 2: TAK-788 120 mg Fed | Part 2: TAK-788 120 mg Fasted | Part 2: TAK-788 160 mg Fed | Part 2: TAK-788 160 mg Fasted
Number analyzed (Participants) | 6 | 6 | 10 | 10
h*ng/mL | 533.8 (272.07) | 525.8 (301.84) | 706.3 (294.61) | 743.0 (462.07)
Statistical Analysis 1: Comparison: Part 2: TAK-788 120 mg Fed vs Part 2: TAK-788 120 mg Fasted; Test type: Equivalence — [test comment as in outcome 5, analysis 2]; Geometric LS Mean Ratio = 1.0153, 90% CI 2-sided [0.8977 to 1.1483]
Statistical Analysis 2: Comparison: Part 2: TAK-788 160 mg Fed vs Part 2: TAK-788 160 mg Fasted; Test type: Equivalence — [test comment as in outcome 5, analysis 2]; Geometric LS Mean Ratio = 0.9506, 90% CI 2-sided [0.8740 to 1.0339]

12. Primary Outcome: Part 3, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-788
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 3: TAK-788 DiC A | Part 3: TAK-788 DiC B
Number analyzed (Participants) | 12 | 12
h*ng/mL | 738.8 (193.06) | 709.5 (262.84)
Statistical Analysis 1: Comparison: Part 3: TAK-788 DiC A vs Part 3: TAK-788 DiC B; Test type: Equivalence — [test comment as in outcome 5, analysis 2]; Geometric LS Mean Ratio = 0.9603, 90% CI 2-sided [0.8861 to 1.0408]

13. Primary Outcome: Part 2, t1/2z: Terminal Disposition Phase Half-life (t1/2z) for TAK-788
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: hour
Arm/Group | Part 2: TAK-788 120 mg Fed | Part 2: TAK-788 120 mg Fasted | Part 2: TAK-788 160 mg Fed | Part 2: TAK-788 160 mg Fasted
Number analyzed (Participants) | 6 | 6 | 10 | 10
hour | 17.17 (2.629) | 17.60 (4.067) | 20.72 (4.827) | 20.62 (6.854)

14. Primary Outcome: Part 3, t1/2z: Terminal Disposition Phase Half-life (t1/2z) for TAK-788
Time Frame: Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: hour
Arm/Group | Part 3: TAK-788 DiC A | Part 3: TAK-788 DiC B
Number analyzed (Participants) | 12 | 12
hour | 16.38 (2.007) | 16.38 (2.858)

15. Secondary Outcome: Part 1, Cmax: Maximum Observed Plasma Concentration for TAK-788 and Its Active Metabolites AP32960 and AP32914
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1 Cohort 1: TAK-788 20 mg | Part 1 Cohort 2: TAK-788 40 mg | Part 1 Cohort 3: TAK-788 80 mg | Part 1 Cohort 4: TAK-788 120 mg | Part 1 Cohort 5: TAK-788 160 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ng/mL
  TAK-788 | 3.22 (0.938) | 7.85 (4.206) | 14.66 (11.649) | 25.81 (9.682) | 52.21 (27.681)
  Metabolite AP32960 | 1.546 (0.4914) | 3.483 (0.8827) | 8.298 (5.5055) | 13.417 (5.5667) | 25.411 (10.7473)
  Metabolite AP32914 | NA (NA) — Data could not be derived since concentration values were below quantifiable limit less than (<) 0.1 ng/mL. | 0.735 (0.2221) | 1.315 (1.0492) | 2.036 (0.6433) | 4.051 (1.8778)

16. Secondary Outcome: Part 1, Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-788 and Its Active Metabolites AP32960 and AP32914
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1 Cohort 1: TAK-788 20 mg | Part 1 Cohort 2: TAK-788 40 mg | Part 1 Cohort 3: TAK-788 80 mg | Part 1 Cohort 4: TAK-788 120 mg | Part 1 Cohort 5: TAK-788 160 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hour
  TAK-788 | 6.0 [2 to 8.08] | 5.0 [4 to 6] | 4.0 [4 to 8] | 6.0 [2 to 6] | 6.0 [4 to 6]
  Metabolite AP32960 | 6.0 [2 to 8.08] | 4.0 [4 to 6] | 4.0 [2 to 6] | 6.0 [6 to 6] | 5.0 [4 to 6]
  Metabolite AP32914 | NA [NA to NA] — Data could not be derived since concentration values were below quantifiable limit < 0.1 ng/mL. | 6.0 [4 to 8] | 4.0 [4 to 8] | 6.0 [6 to 6] | 6.0 [4 to 6]

17. Secondary Outcome: Part 1, AUCt: Area Under the Plasma Concentration-time Curve From Time 0 to Time t for TAK-788 and Its Active Metabolites, AP32960 and AP32914
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1 Cohort 1: TAK-788 20 mg | Part 1 Cohort 2: TAK-788 40 mg | Part 1 Cohort 3: TAK-788 80 mg | Part 1 Cohort 4: TAK-788 120 mg | Part 1 Cohort 5: TAK-788 160 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
h*ng/mL
  TAK-788 | 59.4 (7.07) | 155.2 (112.06) | 250.4 (197.25) | 448.3 (184.43) | 1007.8 (596.14)
  Metabolite AP32960 | 32.7 (6.41) | 74.9 (21.89) | 159.3 (77.04) | 284.0 (125.52) | 538.5 (196.10)
  Metabolite AP32914 | NA (NA) — Data could not be derived since concentration values were below quantifiable limit less than 0.1 ng/mL. | 11.53 (6.092) | 14.59 (11.845) | 31.74 (11.370) | 80.40 (47.696)

18. Secondary Outcome: Part 1, AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-788 and Its Active Metabolites AP32960 and AP32914
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: The PK set included all participants in the safety set who had no major protocol deviations that would have affected the PK analysis and who had sufficient data to calculate PK parameters. The PK analysis population where data at specified time points were available.
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1 Cohort 1: TAK-788 20 mg | Part 1 Cohort 2: TAK-788 40 mg | Part 1 Cohort 3: TAK-788 80 mg | Part 1 Cohort 4: TAK-788 120 mg | Part 1 Cohort 5: TAK-788 160 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
h*ng/mL
  TAK-788 | 63.6 (7.11) | 160.4 (115.57) | 256.9 (203.43) | 456.1 (187.20) | 1017.3 (599.11)
  Metabolite AP32960 | 37.4 (6.23) | 79.8 (22.41) | 165.9 (81.28) | 293.4 (124.35) | 548.0 (198.24)
  Metabolite AP32914: number analyzed (Participants) | 6 | 2 | 5 | 6 | 6
  Metabolite AP32914 | NA (NA) — Data could not be derived since concentration values were below quantifiable limit less than 0.1 ng/mL. | 19.27 (3.111) | 20.34 (12.714) | 34.58 (11.482) | 85.16 (48.623)

19. Secondary Outcome: Part 1, t1/2z: Terminal Disposition Phase Half-life (t1/2z) for TAK-788 and Its Active Metabolites AP32960 and AP32914
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: as for outcome 18
Measure: Geometric Mean (Standard Deviation); unit: hour
Arm/Group | Part 1 Cohort 1: TAK-788 20 mg | Part 1 Cohort 2: TAK-788 40 mg | Part 1 Cohort 3: TAK-788 80 mg | Part 1 Cohort 4: TAK-788 120 mg | Part 1 Cohort 5: TAK-788 160 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hour
  TAK-788 | 18.07 (1.477) | 15.95 (4.593) | 14.25 (4.310) | 18.30 (1.286) | 19.85 (5.464)
  Metabolite AP32960 | 23.96 (3.461) | 21.43 (2.979) | 22.19 (1.137) | 28.93 (5.903) | 29.18 (6.368)
  Metabolite AP32914: number analyzed (Participants) | 6 | 2 | 5 | 6 | 6
  Metabolite AP32914 | NA (NA) — Data could not be derived since concentration values were below quantifiable limit less than 0.1 ng/mL. | 13.75 (3.323) | 12.22 (2.084) | 12.02 (1.162) | 16.09 (4.548)

20. Secondary Outcome: Parts 2 and 3: Number of Participants Reporting One or More TEAEs
Time Frame: Baseline up to 30 days after the last dose of study drug (Day 38) (end of Intervention Period 2)
Population: The safety set included all participants who received any study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Part 3: TAK-788 160 mg DiC A: TAK-788 160 mg, DiC A (reference), orally, under fasted condition, once on Day 1 of Intervention Period 1.
- Part 3: TAK-788 160 mg DiC B: TAK-788 160 mg, DiC B (test), orally, under fasted condition, once, on Day 1 of Intervention Period 1.
Arm/Group | Part 2: TAK-788 120 mg Fed | Part 2: TAK-788 120 mg Fasted | Part 2: TAK-788 160 mg Fed | Part 2: TAK-788 160 mg Fasted | Part 3: TAK-788 160 mg DiC A | Part 3: TAK-788 160 mg DiC B
Number analyzed (Participants) | 6 | 6 | 10 | 10 | 12 | 13
Participants | 3 | 3 | 7 | 5 | 4 | 4

21. Secondary Outcome: Parts 2 and 3: Number of Participants With One or More SAEs
Time Frame: Baseline up to 30 days after the last dose of study drug (Day 38) (end of Intervention Period 2)
Population: The safety set included all participants who received any study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: TAK-788 120 mg Fasted: TAK-788, 120 mg, capsule, orally, once on Day 1 of Intervention Period 1 under fasted conditions (Treatment B).
- Part 2: TAK-788 160 mg Fasted: TAK-788, 160 mg, capsule, orally, once on Day 1 of Intervention Period 1 under fasted conditions (Treatment B).
Arm/Group | Part 2: TAK-788 120 mg Fed | Part 2: TAK-788 120 mg Fasted | Part 2: TAK-788 160 mg Fed | Part 2: TAK-788 160 mg Fasted | Part 3: TAK-788 160 mg DiC A | Part 3: TAK-788 160 mg DiC B
Number analyzed (Participants) | 6 | 6 | 10 | 10 | 12 | 13
Participants | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Parts 2 and 3: Number of Participants With Clinically Significant Abnormal Laboratory Values
Time Frame: Baseline up to 30 days after the last dose of study drug (Day 38) (end of Intervention Period 2)
Population: The safety set included all participants who received any study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: TAK-788 160 mg: TAK-788, 160 mg, capsule, orally, once on Day 1 of Intervention Period 1 under fed conditions with low-fat meal (Treatment A).
Arm/Group | Part 2: TAK-788 120 mg Fed | Part 2: TAK-788 120 mg Fasted | Part 2: TAK-788 160 mg | Part 2: TAK-788 160 mg Fasted | Part 3: TAK-788 160 mg DiC A | Part 3: TAK-788 160 mg DiC B
Number analyzed (Participants) | 6 | 6 | 10 | 10 | 12 | 13
Participants | 0 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Parts 2 and 3: Number of Participants With Clinically Significant Abnormal Vital Signs
Time Frame: Baseline up to 30 days after the last dose of study drug (Day 38) (end of Intervention Period 2)
Population: The safety set included all participants who received any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: TAK-788 120 mg Fed | Part 2: TAK-788 120 mg Fasted | Part 2: TAK-788 160 mg Fed | Part 2: TAK-788 160 mg Fasted | Part 3: TAK-788 160 mg DiC A | Part 3: TAK-788 160 mg DiC B
Number analyzed (Participants) | 6 | 6 | 10 | 10 | 12 | 13
Participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: TEAEs are adverse events that started after the first dose of study drug and no more than 30 days (up to Day 31 in Part 1; Day 38 in Parts 2 and 3 [end of intervention period 2]) after the last dose of study drug
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part 1: Pooled Placebo | Part 1 Cohort 1: TAK-788 20 mg | Part 1 Cohort 2: TAK-788 40 mg | Part 1 Cohort 3: TAK-788 80 mg | Part 1 Cohort 4: TAK-788 120 mg | Part 1 Cohort 5: TAK-788 160 mg | Part 2: TAK-788 120 mg Fed | Part 2: TAK-788 120 mg Fasted | Part 2: TAK-788 160 mg Fed | Part 2: TAK-788 160 mg Fasted | Part 3: TAK-788 DiC A | Part 3: TAK-788 DiC B
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/10 | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/10 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 2/10 | 2/6 | 3/6 | 4/6 | 3/6 | 5/6 | 3/6 | 3/6 | 7/10 | 5/10 | 4/13 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Pooled Placebo (N=10) | Part 1 Cohort 1: TAK-788 20 mg (N=6) | Part 1 Cohort 2: TAK-788 40 mg (N=6) | Part 1 Cohort 3: TAK-788 80 mg (N=6) | Part 1 Cohort 4: TAK-788 120 mg (N=6) | Part 1 Cohort 5: TAK-788 160 mg (N=6) | Part 2: TAK-788 120 mg Fed (N=6) | Part 2: TAK-788 120 mg Fasted (N=6) | Part 2: TAK-788 160 mg Fed (N=10) | Part 2: TAK-788 160 mg Fasted (N=10) | Part 3: TAK-788 DiC A (N=13) | Part 3: TAK-788 DiC B (N=12)
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 3 | 4 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 3 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site phlebitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.

DOCUMENTS (2):
  • Study Protocol (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT03482453/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/53/NCT03482453/SAP_001.pdf